CLINICAL TRIAL: NCT02293980
Title: A Phase 1, Multiple-Dose, Dose-Escalation Trial of PT2385 Tablets, a HIF-2α Inhibitor, in Patients With Advanced Clear Cell Renal Cell Carcinoma
Brief Title: A Phase 1, Dose-Escalation Trial of PT2385 Tablets In Patients With Advanced Clear Cell Renal Cell Carcinoma (MK-3795-001)
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Peloton Therapeutics, Inc., a subsidiary of Merck & Co., Inc. (Rahway, New Jersey USA) (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 3795-001; PT2385-101 (Other: Peloton Study ID); MK-3795-001 (Other: Merck)
Record Dates: First submitted 2014-11-14; First posted 2014-11-19 (Estimated); Last update posted 2024-06-17 (Actual); Status verified 2024-05

CONDITIONS: ccRCC; RCC; Kidney Cancer; Clear Cell Renal Cell Carcinoma; Renal Cell Carcinoma
MeSH Terms: conditions — Kidney Neoplasms; Carcinoma, Renal Cell | interventions — PT2385; endothelial PAS domain-containing protein 1; Nivolumab; cabozantinib; belzutifan

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Part 1: MK-3795 (Experimental): Participants with advanced ccRCC receive MK-3795 at an initial dose level of 100mg orally, twice daily (BID) up to approximately 3 weeks. Dose levels will be escalated to identify the maximum tolerated dose (MTD) and/or Recommended Phase 2 Dose (RP2D) for MK-3795. Each escalated dose will be continued for up to approximately 3 weeks before escalating a dose again until a dose limiting toxicity (DLT) is experienced. Thereafter, participants receive RP2D dose of MK-3795 for up to 2 cycles (each cycle length = 28 days) for up to approximately 1 year. Participants may continue to receive MK-3795 beyond 1 year at the discretion of the Sponsor.
  Interventions: Drug: MK-3795
- Part 2: MK-3795 + Nivolumab + Belzutifan (Experimental): Participants with advanced ccRCC in the expansion phase receive the RP2D of MK-3795 orally in combination with nivolumab 240mg by IV infusion over ~60 minutes every 2 weeks for up to ~1 year (12 cycles; each cycle length = 28 days) or until unequivocal progression or treatment discontinuation, whichever occurs later. As per Amendment 09 (29 March 2024), participants will not receive MK-3795. Participants receive nivolumab 240mg by IV infusion over ~60 minutes every 2 weeks in combination with belzutifan 120 mg once daily (QD) for up to ~1 year (12 cycles; each cycle length = 28 days) or until unequivocal progression or treatment discontinuation, whichever occurs later. If participants experience an adverse event, then nivolumab will be discontinued and participants will continue to receive belzutifan 120 mg QD alone for up to ~1 year (12 cycles; each cycle length = 28 days) or until unequivocal progression or treatment discontinuation, whichever occurs later.
  Interventions: Drug: MK-3795; Drug: Nivolumab; Drug: Bezlutifan
- Part 3: MK-3795 + Cabozantinib (Experimental): Participants with advanced ccRCC in the expansion phase receive the RP2D of MK-3795 in combination with cabozantinib 20mg up to 60mg orally QD for up to approximately 1 year (12 cycles; each cycle length = 28 days) or until unequivocal progression or treatment discontinuation, whichever occurs later.
  Interventions: Drug: MK-3795; Drug: Cabozantinib

INTERVENTIONS:
Drug: MK-3795 — Oral administration
  Other Names: PT2385, PT-2385, HIF-2a, MK-3795
Drug: Nivolumab — IV infusion
  Other Names: Opdivo
  Arms: Part 2: MK-3795 + Nivolumab + Belzutifan
Drug: Cabozantinib — Oral administration
  Other Names: Cabometyx
  Arms: Part 3: MK-3795 + Cabozantinib
Drug: Bezlutifan — Oral administration
  Other Names: MK-6482
  Arms: Part 2: MK-3795 + Nivolumab + Belzutifan

SUMMARY:
PART 1: The primary objective of this study is to identify the maximum tolerated dose (MTD) of MK-3795, formerly called PT2385 and/or the recommended Phase 2 dose (RP2D) of MK-3795 in patients with advanced clear cell renal cell carcinoma (ccRCC).

PART 2: The primary objective of this study is to identify the MTD of MK-3795 up to the RP2D, in combination with nivolumab, in patients with advanced ccRCC.As of Amendment 09 (29 Mar 2024), participants with advanced ccRCC will transition from MK-3795 to belzutifan (MK-6482) in combination with nivolumab or belzutifan alone.

PART 3: The primary objective of this study is to identify the MTD of MK-3795 up to the RP2D, in combination with cabozantinib tablets, in patients with advanced ccRCC.

DETAILED DESCRIPTION:
PART 1: This is a Phase 1, multiple-dose, dose-escalation trial of MK-3795, where patients with advanced ccRCC will be assigned to sequential dose cohorts. Patient safety will be monitored with frequent physical examinations, vital sign measurements, electrocardiograms (ECGs), and hematology and chemistry laboratory studies, and by recording all adverse events (AEs). Blood will be obtained for analysis of the concentration of MK-3795 and to assess biomarkers.

PART 2: This is a Phase 1 trial of MK-3795 in combination with nivolumab, where patients with advanced ccRCC will be assigned to dose cohorts. Patient safety will be monitored with frequent physical examinations, vital sign measurements, ECGs, and hematology and chemistry laboratory studies, and by recording all AEs. Blood will be obtained for analysis of the concentration of MK-3795 and to assess biomarkers. As of Amendment 09 (29 Mar 2024), participants with advanced ccRCC will transition from MK-3795 to belzutifan in combination with nivolumab or belzutifan alone.

PART 3: This is a Phase 1 trial of MK-3795 in combination with cabozantinib tablets, where patients with advanced ccRCC will be assigned to dose cohorts. Patient safety will be monitored with frequent physical examinations, vital sign measurements, ECGs, and hematology and chemistry laboratory studies, and by recording all AEs. Blood will be obtained for analysis of the concentration of MK-3795 and cabozantinb and to assess biomarkers.

ELIGIBILITY:
Inclusion Criteria

PART 1

* Has locally advanced or metastatic clear cell renal cell carcinoma (ccRCC) and has progressed during treatment with at least one prior therapeutic regimen
* Has a life expectancy of ≥ 3 months
* Has adequate organ function
* Able to swallow oral medications

PART 2 - In addition to PART 1

* Received no more than three prior systemic treatment regimens in the advanced or metastatic setting
* Must have received at least one but not more than two prior anti-angiogenic therapy regimens

PART 3 - In addition to PART 1

* Must have received at least one vascular endothelial growth factor receptor (VEGFR) targeting tyrosine kinase inhibitor

Exclusion Criteria

PART 1

* Has a history of untreated brain metastasis or history of leptomeningeal disease or spinal cord compression
* Has failed to recover from the reversible effects of prior anticancer therapy
* Has uncontrolled or poorly controlled hypertension
* Is receiving warfarin anticoagulant therapy or expected to require warfarin
* Has had any major cardiovascular event within 6 months prior to study drug administration
* Has any other clinically significant cardiac, respiratory, or other medical or psychiatric condition that might interfere with participation in the trial or interfere with the interpretation of trial results
* Has had major surgery within 4 weeks before first study drug administration
* Has known human immunodeficiency virus (HIV) infection
* Has an active infection requiring systemic treatment
* Is participating in another therapeutic clinical trial

PART 2 - In addition to PART 1

* Has received prior immunotherapy
* Has any active or recent history of a known or suspected autoimmune disease

PART 3 - In addition to PART 1

* Has gastrointestinal (GI) disorders
* Has any history of congenital long QT syndrome

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 110 (Actual)
Dates: Start 2014-11-25 (Actual); Primary Completion 2017-01-31 (Actual); Study Completion 2026-11-30 (Estimated)

PRIMARY OUTCOMES:
Maximum Tolerated Dose (MTD) | Part 1: 3 Weeks, Part 2: 4 Weeks, Part 3: 4 Weeks
  MTD of MK-3795 will be determined. MTD will be defined as the dose level at which 2 or more participants experience a dose limiting toxicity (DLT) which will be deemed intolerable and the dose level below will be declared the MTD.
Recommended Phase 2 Dose (RP2D) | Part 1: 3 Weeks; Part 2: 4 Weeks, Part 3: 4 Weeks
  The RP2D of MK-3795 will be determined. The RP2D will be determined based on the MTD (or the optimal biological dose (OBD) if the MTD is not identified), the overall safety profile with continued treatment, and pharmacokinetic (PK) profile.

SECONDARY OUTCOMES:
Number of Participants Who Experience an Adverse Event (AE) | Up to approximately 9 years
  An AE is defined as any untoward medical occurrence in a participant administered a study treatment which did not necessarily have to have a causal relationship with this treatment. An AE could be any unfavorable and unintended sign (including an abnormal laboratory finding, for example), symptom, or disease temporally associated with the use of study treatment, whether or not considered related to the study treatment. Any worsening (i.e., any clinically significant adverse change in frequency and/or intensity) of a pre-existing condition that is temporally associated with the use of study treatment, is also an AE. The number of participants who experience an AE will be presented.
Best Response (BOR) per Response Evaluation Criteria In Solid Tumors Version 1.1 (RECIST 1.1) | Up to approximately 1 year
  BOR is the best tumor response recorded up until documentation of progression of disease (PD) or death from any cause, or until the patient withdraws consent. Per RECIST 1.1, PD is defined as ≥20% increase in the sum of diameters of target lesions. In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of ≥5 mm. The appearance of one or more new lesions is also considered PD.
Objective Response Rate (ORR) per RECIST 1.1 | Up to approximately 1 year
  ORR is defined as the percentage of participants who have a Complete Response (CR: Disappearance of all target lesions) or a Partial Response (PR: At least a 30% decrease in the sum of diameters of target lesions) per RECIST 1.1. The percentage of participants who experience a CR or PR based on RECIST 1.1 will be presented.
Progression-Free Survival (PFS) per RECIST 1.1 | Up to approximately 9 years
  PFS is defined as the time from the first dose of MK-3795 to the first documented progressive disease (PD) or death due to any cause, whichever occurs first. Per RECIST 1.1, PD is defined as ≥20% increase in the sum of diameters of target lesions. In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of ≥5 mm. The appearance of one or more new lesions is also considered PD.
Duration of Response (DOR) per RECIST 1.1 | Up to approximately 1 year
  For participants who demonstrate a confirmed Complete Response (CR: Disappearance of all target lesions) or confirmed Partial Response (PR: At least a 30% decrease in the sum of diameters of target lesions) per RECIST 1.1, DOR is defined as the time from first documented evidence of CR or PR until progressive disease (PD) or death. Per RECIST 1.1, PD was defined as at least a 20% increase in the sum of diameters of target lesions. In addition to the relative increase of 20%, the sum must also have demonstrated an absolute increase of at least 5 mm. The appearance of one or more new lesions was also considered PD. The median DOR will be presented.
Clinical Benefit Rate (CBR) per RECIST 1.1 | Up to approximately 1 year
  CBR is defined as the percentage of participants who achieve clinical benefit. Clinical benefit is defined as a best response of CR (Disappearance of all target lesions), PR (At least a 30% decrease in the sum of diameters of target lesions) or stable disease (SD: Neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for progressive disease [PD: At least a 20% increase in the sum of diameters of target lesions and an absolute increase of at least 5 mm. The appearance of one or more new lesions is also considered PD.]).
Maximum concentration (Cmax) of Study Treatment | At designated timepoints (up to 106 days)
  Blood samples will be collected at designated timepoints for the determination of Cmax. Cmax was defined as the maximum concentration of study treatment is reached.
Time to Maximum Concentration (Tmax) of Study Treatment | At designated timepoints (up to 106 days)
  Blood samples will be collected at designated timepoints the determination of Tmax. Tmax is defined as the time to the maximum concentration of study treatment reached.
Terminal half-life (t½λz) of Study Treatment | At designated timepoints (up to 106 days)
  Blood samples will be collected at designated timepoints for the determination of (t½λz). (t½λz) is defined as the time required for the plasma concentration of study drug to decrease 50% in the final stage of its elimination.
Area Under the Concentration-Time Curve From 0 to Infinity (AUC0-inf) of Study Treatment | At designated timepoints (up to 106 days)
  Blood samples will be collected at designated timepoints for the determination of AUC0-inf. AUC0-inf is the area under the serum concentration-time curve from time zero to infinity.
Area Under the Concentration-Time Curve From 0 to Inf Extrapolated (AUC0-inf Extrap) of Study Treatment | At designated timepoints (up to 106 days)
  Blood samples were collected at designated timepoints for the determination of AUC0-inf extrapolated. AUC0-inf extrapolated is a measure of mean concentration in serum from time zero to infinity.
Area Under the Concentration-Time Curve From 0 to 12 Hours (AUC0-12) of Study Treatment | At designated timepoints (up to 106 days)
  Blood samples were collected at designated timepoints for the determination of AUC0-12. AUC0-12 is a measure of mean concentration in serum from time zero to 12 hours.
Area Under the Plasma Concentration-time Curve From Time 0 to Last (AUC0-last) of Study Treatment | At designated timepoints (up to 106 days)
  Blood samples were collected at designated timepoints for the determination of AUC0-last. AUC0-last is a measure of mean concentration in serum from time zero to last measurable concentration.
Apparent Volume of Distribution (Vz/F) of Study Treatment | At designated timepoints (up to 106 days)
  Blood samples were collected at designated timepoints for the determination of Vz/F. Vz/F is a the volume of study drug that would need to be uniformly distributed to produce desired serum concentration. F is the fraction of the dose absorbed.
Apparent Clearance (CL/F) of Study Treatment | At designated timepoints (up to 106 days)
  Blood samples were collected at designated timepoints for the determination of CL/F. CL/F is a the volume of plasma from which study drug was eliminated per unit time. F is the fraction of the dose absorbed.
Accumulation Ratio (RAC) | At designated timepoints (up to 106 days)
  Blood samples were collected at designated timepoints for the determination of RAC. RAC is calculated as AUC0-12 at steady state divided by AUC0-12 after first dose.
Mean Plasma Concentration of Erythropoietin (EPO) Level | At designated timepoints (up to 106 days)
  Blood samples will be collected at designated timepoints to measure EPO level. The mean concentration of EPO level will be reported.
Mean Plasma Concentration of Plasminogen Activator Inhibitor 1 (PAI-1) Level | At designated timepoints (up to 106 days)
  Blood samples will be collected at designated timepoints to measure PAI-1 level. The mean concentration of PAI-1 level will be reported.
Mean Plasma Concentration of Insulin Growth Factor Binding Protein 3 (IGFBP3) Level | At designated timepoints (up to 106 days)
  Blood samples will be collected at designated timepoints to measure IGFBP3 level. The mean concentration of IGFBP3 level will be reported.
Mean Plasma Concentration of Vascular Endothelial Growth Factor A (VEGFa) Level | At designated timepoints (up to 106 days)
  Blood samples will be collected at designated timepoints to measure VEGFa level. The mean concentration of VEGFa level will be reported.
Percent Change from Baseline in the EPO Level | Baseline and up to approximately Week 16
  Blood samples will be collected at designated timepoints to measure EPO level. The percent change from baseline in EPO level up to approximately Week 16 will be reported.
Percent Change from Baseline in the PAI-1 Level | Baseline and up to approximately Week 16
  Blood samples will be collected at designated timepoints to measure PAI-1 level. The percent change from baseline in PAI-1 level up to approximately Week 16 will be reported.
Percent Change from Baseline in the IGFBP3 Level | Baseline and up to approximately Week 16
  Blood samples will be collected at designated timepoints to measure IGFBP3 level. The percent change from baseline in IGFBP3 level up to approximately Week 16 will be reported.
Percent Change from Baseline in the VEGFa | Baseline and up to approximately Week 16
  Blood samples will be collected at designated timepoints to measure VEGFa level. The percent change from baseline in VEGFa level up to approximately Week 16 will be reported.
Antitumor Activity | Baseline, at Week 6 and every 9 Weeks thereafter up to approximately 1 year
  Antitumor activity will be assessed by non-contrast or contrast computerized tomography (CT) or magnetic resonance imaging (MRI) at baseline, during Week 6, and every 9 weeks thereafter up to approximately 1 year.

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC
Locations (25):
- United States (25):
  - Cedars-Sinai Medical Center, Los Angeles, California
  - University of Colorado Cancer Center, Aurora, Colorado
  - Yale School of Medicine, New Haven, Connecticut
  - University of Miami - Sylvester Comprehensive Cancer Center, Miami, Florida
  - Emory University Winship Cancer Institue, Atlanta, Georgia
  - Rush University Medical Center, Chicago, Illinois
  - Indiana University Simon Cancer Center, Indianapolis, Indiana
  - University of Maryland - Greenebaum Cancer Center, Baltimore, Maryland
  - Massachusetts General Hospital - Cancer Center, Boston, Massachusetts
  - Beth Israel Deconess Medical Center, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Barbara Ann Karmanos Cancer Institute, Detroit, Michigan
  - Mount Sinai Heath System, New York, New York
  - Cleveland Clinic, Cleveland, Ohio
  - The Ohio State University, Columbus, Ohio
  - Fox Chase Cancer Center, Philadelphia, Pennsylvania
  - University of Pittsburg Medical Center, Pittsburgh, Pennsylvania
  - The West Clinic, Germantown, Tennessee
  - Tennessee Oncology, Nashville, Tennessee
  - Vanderbilt Medical Center, Nashville, Tennessee
  - UT Southwestern Medical Center, Dallas, Texas
  - Virginia Cancer Specialists, Fairfax, Virginia
  - Swedish Cancer Institute, Seattle, Washington
  - University of Washington, Seattle, Washington
  - Medical College of Wisconsin, Milwaukee, Wisconsin

IPD SHARING:
Plan to Share IPD: Yes
http://engagezone.msd.com/doc/ProcedureAccessClinicalTrialData.pdf
URL: http://engagezone.msd.com/ds_documentation.php

REFERENCES:
- [Derived] Courtney KD, Infante JR, Lam ET, Figlin RA, Rini BI, Brugarolas J, Zojwalla NJ, Lowe AM, Wang K, Wallace EM, Josey JA, Choueiri TK. Phase I Dose-Escalation Trial of PT2385, a First-in-Class Hypoxia-Inducible Factor-2alpha Antagonist in Patients With Previously Treated Advanced Clear Cell Renal Cell Carcinoma. J Clin Oncol. 2018 Mar 20;36(9):867-874. doi: 10.1200/JCO.2017.74.2627. Epub 2017 Dec 19. PMID 29257710
- See also: Merck Clinical Trials Information — https://www.merckclinicaltrials.com/